CLINICAL TRIAL: NCT00243334
Title: Improving Safety and Quality With Outpatient Order Entry
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Tejal Gandhi, Associate Professor, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 5R01HS015226-02 (AHRQ)
Record Dates: First submitted 2005-10-21; First posted 2005-10-24 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Ambulatory Care Information Systems; Clinical Decision Support Systems
Keywords: Ambulatory Care Information Systems; Clinical Decision Support Systems; Medication Systems; Medication Errors; Reminder Systems; Drug Monitoring; Preventive Health Services; Time and Motion Studies; Efficiency; Cost-Benefit Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Decision Support integrated with Order Entry
  Interventions: Other: Integration of advanced clinical decision support with ambulatory computerized physician order entry
- 2 (No Intervention): Decision Support Only (not integrated with order entry)

INTERVENTIONS:
Other: Integration of advanced clinical decision support with ambulatory computerized physician order entry — Actiobable Reminders related to medication monitoring, preventive care and chronic disease management, and test result follow-up are administered either during the visit or between visits.
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the impact of integrating ambulatory computerized physician order entry (ACPOE) and advanced clinical decision support systems (CDSS) on safety and quality domains in the ambulatory setting, including: a) medication monitoring, b) preventive care and chronic disease management, and c) test result follow-up. In addition we will evaluate the impact on organizational efficiency, physician workflow and satisfaction, and perform a cost-benefit analysis. We hypothesize that the value of ACPOE integrated with advanced CSDSS lies in improved medication safety and guideline compliance, but also improved efficiencies for the provider and the health-care system.

DETAILED DESCRIPTION:
Quality gaps that are relevant to the ambulatory setting include a high incidence of adverse drug events and lack of compliance to established guidelines for preventive care, chronic disease management and test result follow-up. Clinical decision support systems (CDSS) and ambulatory computerized physician order entry (ACPOE) have been touted as powerful interventions to address these concerns. However, doubts exist about the efficacy of these systems in the ambulatory setting, especially when they exist in isolation. Also, despite the evidence of the impact of inpatient CPOE, the impact of ACPOE has not been well studied. Moreover, the adoption of CDSS and ACPOE systems is slow, and their value proposition remains uncertain.

Tightly integrating CDSS with ACPOE serves as a promising strategy to improve quality and efficiency in the ambulatory setting by facilitating physician action. When ACPOE is linked with CDSS, clinicians can be prompted at various points during their workflow about the desirable course of action and simultaneously be given the opportunity to execute the action (by ordering it) with minimal effort. We hypothesize that the value of ACPOE integrated with advanced CSDSS lies in improved medication safety and guideline compliance, but also improved efficiencies for the provider and the health-care system. We further hypothesize that the value added by these systems overall out weights their costs. This study will evaluate the impact of integrating ACPOE with advanced CDSS on important safety and quality domains in the ambulatory setting using randomized controlled trials. In addition, we will evaluate the impact on organizational efficiency, physician workflow and satisfaction, and perform a cost-benefit analysis.

There are 2 interventions periods. During Intervention Period 1, a randomized selection of clinics (Arm 1) will receive basic order entry without integrated decision support (i.e. no intervention) while another randomized selection of clinics (Arm 2) receive order entry integrated with decision support in the form of delivery of reminders and alerts during a clinical encounter (Intervention A). During Intervention Period 2, Arm 2 clinics will continue to receive Intervention A. However, Arm 1 clinics receive Intervention A plus additional decision support delivered in between clinic encounters (Intervention B).

Comparisons:

We will evaluate the impact of Intervention A (during visit) and intervention B (between visits) in 2 clustered randomized controlled trials, giving us accurate estimates of their individual efficacies. This is particularly important because these findings will highlight the relative value of these 2 different modes of decision support and inform organizations and vendors about how to invest their development resources. We also will be able to evaluate the combined impact of interventions A and B (between visits) by comparing the outcome in Arm 2 across the 2 intervention periods while simultaneously controlling for any secular trends (as observed in Arm 1 across the 2 intervention periods). All clinics, regardless of randomization status, will have access to at least one intervention during study period.

ELIGIBILITY:
Inclusion Criteria:

* All physicians in on-site and satellite adult outpatient clinics with the Brigham and Women's Hospital and Massachusetts General Hospital

Exclusion Criteria:

* Study clinics must have adopted our electronic health record system, the Longitudinal Medical Record, for at least 24 months and must have implemented the basic version of the internally-developed lab order entry module.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-12 (Actual); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Whether an instance that requires ordering of an appropriate laboratory test or medication or other appropriate monitoring action (based on guidelines and electronic clinical data) is associated with appr opriate action. | Within 14 days of a patient visit or 28 days of the arrival of a test result
Whether the incidence of a particular abnormal result (based on guidelines and electronic clinical data) was associated with the appropriate follow-up. | Varies by major test type
Whether a test ordered does not get performed. | Varies by major test type

SECONDARY OUTCOMES:
The time to appropriate action following the firing of a reminder. | Within 14 days of the reminder firing
The time to appropriate monitoring action following the arrival of the index lab result. | Within 28 days of lab result
The time to appropriate follow-up following a particular abnormal result. | Within 28 days of the result

CONTACTS AND LOCATIONS:
Overall Officials: Tejal K Gandhi, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Partners HealthCare System, Inc., Boston, Massachusetts, United States